CLINICAL TRIAL: NCT01994863
Title: An Open-labeled, Randomised, Controlled, Comparative, Cross-over Study Investigating the Safety and Performance of a New 1-piece Ostomy Product Compared to Standard Care 1-piece in Subjects With Ileostomy
Brief Title: Safety and Performance Investigation of a New 1-piece Ostomy Product Compared to Standard of Care 1-piece in Subjects With Ileostomy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Problems with product performance
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CP224
Record Dates: First submitted 2013-02-26; First posted 2013-11-26 (Estimated); Results first posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Ileostomy - Stoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- First Coloplast Test product; then Standard Care (see below) (Experimental): The subjects are randomised to test Coloplast Test product first and thereafter test Standard Care.
  Standard Care is a collection of three different already marketed 1-piece flat ostomy appliances. These are Coloplast Sensura 1-piece; Hollister: Moderma 1-piece and B.Braun Flexima 1-piece.
  The three Standard Care products were tested in a 1:1:1 randomisation.
  Interventions: Device: Coloplast Test product; Device: Standard Care
- First Standard Care (see below); Then coloplast test product (Experimental): The subjects are randomised to test Standard care first and thereafter test Coloplast test product.
  Standard Care is a collection of three different already marketed 1-piece flat ostomy appliances. These are Coloplast Sensura 1-piece; Hollister: Moderma 1-piece and B.Braun Flexima 1-piece.
  The three Standard Care products were tested in a 1:1:1 randomisation.
  Interventions: Device: Coloplast Test product; Device: Standard Care

INTERVENTIONS:
Device: Coloplast Test product — Coloplast test product is a newly developed 1-piece ostomy appliance
  Other Names: Coloplast 1-piece test product
Device: Standard Care — Standard care consists of three already marketed 1-piece ostomy products
  Coloplast SenSura Hollister Moderma/Moderma Flex B.Braun Flexima/Softima
  Other Names: Coloplast SenSura; Hollister Moderma/Moderma Flex; B.Braun Flexima/Softima

SUMMARY:
The objective of the investigation is to document New Mio 1-piece is non-inferior (no worse) in reducing leakage (4-point scale) compared to Standard of Care.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent
2. Be at least 18 years of age and have full legal capacity
3. Be able to handle the appliance themselves or with help from caregiver (e.g. spouse)
4. Have an ileostomy with a diameter between 15 and 45 mm
5. Have had their ostomy for at least three months
6. Currently use a 1-piece flat product with open bag
7. Use minimum 1 product every second day.
8. Be suitable for participation in the investigation and for using a standard adhesive, flat base plate
9. Must use custom cut product
10. Accept to test two 1-piece products within the study

Exclusion Criteria:

1. Use irrigation during the study (flush the stoma with water)
2. Currently receiving or have within the past 2 months received radio- and/or chemotherapy
3. Currently receiving or have within the past month received systemic steroid or local treatment in the peristomal area
4. Are pregnant or breastfeeding
5. Participating in other interventional clinical investigations or have previously participated in this investigation
6. Has more than three days wear time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Carter, MSc, Study Director — Coloplast A/S
Locations (1):
- QPS Netherland B.V., Groningen, Netherlands

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: "Not completed" includes those who did not complete the entire period (those that did not try all products within the period) and then continued to next period, if relevant.
Groups:
- First Coloplast Test Product; Then Standard Care (See Below): The subjects are randomised to test Coloplast Test product first and thereafter test Standard Care.
  Standard Care is a collection of three different already marketed 1-piece flat ostomy appliances. These are Coloplast Sensura 1-piece; Hollister: Moderma 1-piece and B.Braun Flexima 1-piece.
  The three Standard Care products were tested in a 1:1:1 randomisation.
  Coloplast Test product: Coloplast test product is a newly developed 1-piece ostomy appliance
  Standard Care: Standard care consists of three already marketed 1-piece ostomy products
  Coloplast SenSura Hollister Moderma/Moderma Flex B.Braun Flexima/Softima
- First Standard Care (See Below); Then Coloplast Test Product: The subjects are randomised to test Standard care first and thereafter test Coloplast test product.
  Standard Care is a collection of three different already marketed 1-piece flat ostomy appliances. These are Coloplast Sensura 1-piece; Hollister: Moderma 1-piece and B.Braun Flexima 1-piece.
  The three Standard Care products were tested in a 1:1:1 randomisation.
  Coloplast Test product: Coloplast test product is a newly developed 1-piece ostomy appliance
  Standard Care: Standard care consists of three already marketed 1-piece ostomy products
  Coloplast SenSura Hollister Moderma/Moderma Flex B.Braun Flexima/Softima
Period: Period 1
Arm/Group | First Coloplast Test Product; Then Standard Care (See Below) | First Standard Care (See Below); Then Coloplast Test Product
Started | 11 | 12
Completed | 4 | 9
Not Completed | 7 | 3
Not completed — Adverse Event | 4 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Trial stopped by sponsor | 1 | 3
Not completed — Lack of Efficacy | 1 | 0
Period: Period 2
Arm/Group | First Coloplast Test Product; Then Standard Care (See Below) | First Standard Care (See Below); Then Coloplast Test Product
Started | 8 | 9
Completed | 7 | 5
Not Completed | 1 | 4
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 13
Region of Enrollment [Number; unit: participants]
  Netherlands | 17
  France | 6

OUTCOME MEASURES:

1. Primary Outcome: Leakage
Description: The percentage of baseplates with no leakage/seeping under the baseplate was measured. Leakage/seeping under the baseplate was assessed after each baseplate change.
Time Frame: 14+/-3 days per product
Population: Intention-to-treat population
Measure: Number; unit: percentage of baseplates with no leakage
Units Other Than Participants: Baseplates
Arm/Group | Coloplast Test Product | Standard Care
Number analyzed (Participants) | 20 | 19
Number analyzed (Baseplates) | 145 | 180
percentage of baseplates with no leakage | 50 | 77

ADVERSE EVENTS:
Arm/Group | Coloplast Test Product | Standard Care
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 8/20 | 6/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coloplast Test Product (N=20) | Standard Care (N=20)
Peristomal skin problem/pain/itching (Skin and subcutaneous tissue disorders) | 8 (9) | 6 (6) — Possibly related to the product

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days